CLINICAL TRIAL: NCT01097421
Title: Influence of Pramipexole Extended Release on Medication Adherence in Real Life Care of Parkinson's Disease
Brief Title: Influence of Pramipexole Extended Release on Medication Adherence in Parkinson´s Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.674
Record Dates: First submitted 2010-03-25; First posted 2010-04-01 (Estimated); Results first posted 2012-11-26 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patient with parkinsons disease
  Interventions: Drug: Pramipexole Extended Release

INTERVENTIONS:
Drug: Pramipexole Extended Release

SUMMARY:
This is an open-label, prospective post marketing surveillance study to be performed in Sweden. Only data of patients idiopathic PD should be documented, in whom the treating physician plans to initiate a pharmacotherapy with PPX ER independent of this observational study. The questionnaires (Morisky Medication Adherence Measure, patient preference scale, CGI-I, PGI-I) will be used to document routine care in a standardized way and thus ensure high validity of the observational data. As the degree medication adherence of patients is routinely evaluated by their physicians, as is patient preference and possible symptom improvement after initiation of a new therapy, the patient questionnaires will be used to standardise medical routine care and to ensure validity of observational data.

ELIGIBILITY:
Inclusion criteria:

1. Patients suffering from idiopathic PD who before inclusion into the observation had been planned to be treated with PPX ER according to the SP, and where decision of treatment was made independently of the patients¿ inclusion into this observational study
2. Stable dose of PPX IR for at least 4 weeks before inclusion into the observation
3. Male or female PD patients aged at least 30
4. Ability to reliably complete self-rating scales (Morisky Medication Adherence Measure, patient preference scale) according to the physician¿s judgement
5. Written informed consent by the patient for study participation.

Exclusion criteria:

1. Patients who are not able to understand the questionnaires (e.g. due to mental impairment or language problems) according to the physician¿s judgement.
2. Any contraindications against PPX ER according to the Summary of Product Characteristics (SPC).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: specialist care
Sampling Method: Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2010-03; Primary Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 328 patients entered and treated with a documented baseline observation in this study.
Pre-assignment Details: This was an open-label, prospective, non-controlled, non-interventional observational, post marketing surveillance study.
Groups:
- Pramipexole Extended Release: individual doses planned in the range of 0.26 mg (0.375 mg of salt) to 3.15 mg (4.5 mg of salt) of base per day
Period: Overall Study
Arm/Group | Pramipexole Extended Release
Started | 328
Completed | 314
Not Completed | 14
Not completed — Adverse Event | 8
Not completed — Protocol Violation | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS)
Arm/Group | Pramipexole Extended Release
Number analyzed (Participants) | 326
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116
  Male | 210

OUTCOME MEASURES:

1. Primary Outcome: Patients With a Score of 4 in Morisky Scale After 8-12 Weeks of Treatment
Description: Morisky scale: 4 Yes/No Questions: Do you ever forget to take your medicine? Are you careless at times about taking your medicine? When you feel better do you sometimes stop taking your medicine? Sometimes if you feel worse when you take the medicine, do you stop taking it? Score one point for every NO: 0-1 points = low adherence, 2-3 points = moderate, 4 points = high adherence Confidence interval computed using the Clopper-Pearson (exact) method.
Time Frame: 8-12 weeks
Population: Full Analysis Set (FAS) defined as all patients who had taken at least one dose of the investigational medicinal product (IMP) and had a post-baseline assessment.
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Pramipexole Extended Release
Number analyzed (Participants) | 326
Percent | 75.2 ((70.1, 79.8)) [70.1 to 79.8]

2. Primary Outcome: Level of Adherence
Description: Points on Morisky scale
Time Frame: 8-12 weeks
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Pramipexole Extended Release
Number analyzed (Participants) | 326
Participants
  Low Adherence | 4
  Moderate Adherence | 77
  High Adherence | 245

3. Secondary Outcome: Patient Preference
Description: Patients were asked about their preference regarding frequency of intake (once daily or three times daily)
Time Frame: 8-12 weeks
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Pramipexole Extended Release
Number analyzed (Participants) | 326
Participants
  Once daily intake | 284
  Three times daily intake | 18
  No difference | 24

4. Secondary Outcome: Adverse Events (AE) Considered Related to Observed Medication
Description: Some patients had not related AEs as well as related AEs.
Time Frame: 8-12 weeks
Population: Safety Analysis Set (SAS) defined as all treated patients with a documented baseline observation.
Measure: Number; unit: Patients
Arm/Group | Pramipexole Extended Release
Number analyzed (Participants) | 328
Patients
  related | 20
  not related | 21
  total AE - related and not related | 39

5. Secondary Outcome: Pramipexole (PPX) Dose
Description: mean Pramipexole (PPX) dose
Time Frame: pre-treatment and after 8-12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: mg/24 hr
Arm/Group | Pramipexole Extended Release
Number analyzed (Participants) | 326
mg/24 hr
  pre-treatment immediate release dose | 1.07 (0.73)
  extended release dose at final observation | 1.05 (0.75)

6. Secondary Outcome: Clinical Global Impressions (CGI)
Description: Clinical Global Impression (CGI) scale at final visit
Time Frame: 8-12 weeks
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Pramipexole Extended Release
Number analyzed (Participants) | 326
Participants
  Very much improved | 0
  Much improved | 38
  Minimally improved | 106
  No change | 149
  Minimally worse | 26
  Much worse | 7
  Very much worse | 0

7. Secondary Outcome: Patients Global Impressions (PGI)
Description: Assessed by asking the patient at the final visit which alternative described how they had felt during the last 7 days as compared to how they felt at the baseline observation.
Time Frame: 8-12 weeks
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Pramipexole Extended Release
Number analyzed (Participants) | 326
Participants
  Very much improved | 3
  Much improved | 45
  Minimally improved | 91
  No change | 138
  Minimally worse | 39
  Much worse | 9
  Very much worse | 1

ADVERSE EVENTS:
Time Frame: 8-12 weeks
Arm/Group | Pramipexole Extended Release
Serious Adverse Events (participants affected / at risk) | 3/328
Other Adverse Events (participants affected / at risk) | 0/328
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole Extended Release (N=328)
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Sudden death (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.